CLINICAL TRIAL: NCT00443911
Title: Rheohemapheresis and Lutein Supplementation (Xantophyll Carotenoid) in the Non-Exsudative Form of Age-Related Macular Degeneration
Brief Title: Rheohemapheresis and Lutein Supplementation in the Non-Exsudative Form of Age-Related Macular Degeneration
Acronym: ReLux-AMD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Prof.Dr. Susanne Binder, Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery
Other Study IDs: LBI-06-053-0406
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macular degeneration, rheopheresis, lutein
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Age-related macular degeneration is one of the major causes of blindness in the western world. There is an exsudative and a non-exsudative form of age-related macular degeneration.Most studies concentrate on the exsudative form. In the non-exsudative form the policy is generally watch and see, but patients are at risk to develop an exsudative form. So far, the only accepted therapy to reach stable disease in the non-exsudative form is high-dose supplementation of antioxidants. Another approach to improve visual acuity in patients with non-exsudative form of macular degeneration is rheohemapheresis treatment, an extracorporeal therapy where plasma is separated from blood cells. By the use of a hollow fiber filter plasma is depleted of high molecular weight proteins and reinfused. Others report describe the supplementation of lutein (a vitamin A derivative) as possible treatment option. However, none of the studies have yet examined a combination of rheohemapheresis and lutein supplementation.

DETAILED DESCRIPTION:
Rheohemapheresis will be performed in 5 cycles. One cycle consists of 2 rheohemapheresis treatments on day 1 and day 4. A cycle lasts for 4 weeks and will be repeated every fourth week. During each treatment > 75% to 100% of patients total plasma volume has to be filtered.General medical reviews, ETDRS and Radner visual acuity assessment, ophthalmologic examinations, ocular imaging with OCT 3, autofluorescein imaging and infrared imaging, multifocal ERG, ocular echography, and blood examinations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Study eye with non-exsudative AMD AREDS II - III

  * with > 10 large soft, and / or confluent drusen within 3000 nm of the foveal centre
  * and a best corrected visual acuity of 0.06 - 1.0 using ETDRS charts (letter score of 3 to 50 letters)
  * with / without geographic atrophy less than 3 disc diameters within 3000 nm of the foveal centre ´. with / without serous pigment epithelial detachment without clearly identifiable neovascularisation
* Patients must have elevated baseline concentrations of at least one of the rheologic parameters (serum cholesterol level > 200 mg/dL, fibrinogen level > 390 mg/dL, or plasmaviscosity > 1.6 mPa*s)
* Men or women aged between 50 - 99 years.

Exclusion Criteria:

* Study eye with exsudative AMD
* Study eye with concomitant retinal or choroidal disorder other than AMD
* Study eye with significant central lens opacities and / or conditions that limit the view of the fundus
* poor general condition
* hematocrit < 30%
* coagulation disorders (incl. marcoumar therapy)
* significant cardiac problems ( > NYHA II)
* history (< 12 months) of cardiac infarction
* uncontrolled arterial hypertension
* recent history (< 3 months) of cerebral vascular infarction
* cerebrovascular disease IV
* uncontrolled diabetes
* insufficient antecubital venous access
* lutein supplementation within the last 3 months
* weight < 45 kg
* hemato-oncological disorder
* Patients who are unwilling to adhere to visit examination schedules

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-exudative AMD
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Katharina E Kubista, MD, Principal Investigator — LBI
Locations (1):
- Rudolf Foundation Clinic, Department of Ophthalmology, Vienna, Vienna, Austria